CLINICAL TRIAL: NCT01160029
Title: RANDOMIZED, 2-WAY CROSSOVER, BIOEQUIVALENCE STUDY OF NATEGLINIDE 120 mg TABLET AND STARLIX@ ADMINISTERED AS 1 x 120 mg TABLET IN HEALTHY SUBJECTS UNDER FASTING CONDITIONS
Brief Title: Bioequivalence Study of Nateglinide Tablets 120 mg of Dr. Reddy's Laboratories Limited Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice president- Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40332
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2004-09

CONDITIONS: Healthy
MeSH Terms: interventions — Nateglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nateglinide (Experimental): Nateglinide Tablets 120 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Nateglinide
- Starlix (Active Comparator): Starlix Tablets 120 mg of Novartis
  Interventions: Drug: Nateglinide

INTERVENTIONS:
Drug: Nateglinide — Nateglinide Tablets 120 mg
  Other Names: Starlix tablets 120 mg

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of nateglinide 120 mg tablet (test) versus Starlix ® (reference), administered as 1 x 120 mg tablet under fed conditions.

DETAILED DESCRIPTION:
Single center, bioequivalence, open-label, randomized, 2-way crossover study. 54 + 4 healthy adult male or female, smokers and/or non-smokers. Single oral dose (1 x 120 mg) in each period with a washout of at least 7 days between doses. Dosing with 240 ml of glucose solution (25%).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, smoker or non-smoker, 18 years of age and older.
* Capable of consent

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* BMI>30kg/m2
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol),
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, nateglinide, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption or hormonal contraceptives.
* Difficulty to swallow study medication.
* Smoking more than 10 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptive) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Patients affected by Type 1 diabetes or diabetic ketoacidosis (this last condition should be treated with insulin).
* Breast-feeding.
* Positive serum pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner within 14 days prior to study drug administration. Acceptable methods of contraception:
* condom + spermicide;
* diaphragm + spermicide;
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration);
* hormonal contraceptives (starting at least 4 weeks prior to study drug administration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Pizarro, MD, Principal Investigator — SFBC International, SFBC Miami, Inc. 11190 Biscayne Blvd.Miami, Fl 33181, USA